CLINICAL TRIAL: NCT02740647
Title: The Efficiency of Postoperative Antibiotics in Orthognathic Surgery: A Prospective, Randomized, Double-blind, Placebo-controlled Clinical Trial
Brief Title: The Efficiency of Postoperative Antibiotics in Orthognathic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Baruch Padeh Medical Center, Poriya (Other Government)
Responsible Party: Principal Investigator, Yasmen Ghantous, Dr., The Baruch Padeh Medical Center, Poriya
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0077-14.CTIL
Record Dates: First submitted 2016-03-20; First posted 2016-04-15 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Asymptomatic Diseases
MeSH Terms: conditions — Asymptomatic Diseases | interventions — Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention group (Experimental): Intervention group will be getting intra-venous1GR Amoxicillin Clavulanate 3 times a day for 5 days post surgery.
  Interventions: Drug: Amoxicillin Clavulanate
- Control group (Placebo Comparator): the Control group will be getting intra-venous Placebo (0.9% 50 ml of sodium chloride) for 5 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Amoxicillin Clavulanate — getting intra-venous1GR Amoxicillin Clavulanate 3 times a day for 5 days post surgery
  Other Names: Augmantin
  Arms: Intervention group
Drug: Placebo — 50 ml of 0.9% sodium chloride three times a day
  Arms: Control group

SUMMARY:
Orthognathic surgery is the state of art of the maxillofacial surgery, it fix and normalize facial abnormalities and create a harmony between the different tissues compounding the face (bone, soft tissue and dental structures). It is a common procedure and it is done in order to correct a dentofacial and skeletal deformities.

There is an inevitable risk of complications with this type of surgery. While postoperative infections are the most common complication (2% to 33.4%).

preoperative administration of antibiotics have been proven to be effective in reducing the postoperative infection rate, while, the quality of the currently available literature in prescribing continues postoperative antibiotics is questionable and there is still no consensus on its efficacy.

Unwise administration of antibiotics may cause several unwanted side effects such as gastrointestinal symptoms, allergy reactions, high costs, etc… while the most worrisome side effect is a bacterial resentence.

The objective of this study is to investigate the efficacy of postoperative antibiotics. And will try to state a consensus in prescribing postoperative antibiotics. By conducting a prospective, randomized, double-blind, placebo-controlled study, that will explore and analyze the efficacy of postoperative administration of Amoxicillin Clavulanate versus placebo in reducing the rate of postoperative infections in 60 healthy patients.

DETAILED DESCRIPTION:
The first Orthographic operation was carried out in 1849, for the correction of malocclusions, in the United States of America. Back then, this surgery was merely a mandibular operation and was called Hullihen's procedure done by general surgeons. However, the first cooperation between surgeons and orthodontists in the evolution of the early orthognathic surgery was cradled in St. Louis by the orthodontist Edward Angle (1898) and the surgeon Vilray Blair (1906). During the 19th orthognathic surgery underwent minor improvements, never the less, not until the beginning of the 1950s, when orthognathic surgery was deemed as a true specialty had its origins, which led to tremendous success all over the world. Nowadays, orthognathic surgery is performed not only for correcting dental and skeletal deformities, but also is conducted as a treatment of various congenital and cranio-facial syndromes, such as Crouzon syndrome, Treacher syndrome and Apert's syndrome.

However, orthognathic surgery is not an innocent procedure, since it contains several complications. Pain, swelling, neurosensory deficits and post operative infections are the most common complications. While postoperative infection is the most common one, with a 2% to 33.4% percentage of occurrences. Postoperative infections increase the mortality rate of orthognathic procedure and may create a challenge for the surgeon and the medical staff, thus, reducing its prevalence is critical issue in defining the success of this unique procedure.

Preoperative prophylaxis has been proven as an efficient in decreasing the rate of postoperative infections in orthognathic surgery.

While the current literature regarding the efficacy of postoperative antibiotics questionable and there is still no consensus on its efficacy.

This study is a prospective, randomized, double-blind, placebo-controlled study that will investigate the efficacy of postoperative antibiotics. And will try to state a consensus in prescribing postoperative antibiotics.

Objectives and Goals of the study:

The main goal of the present study is to evaluate the efficacy of post operative antibiotics in decreasing the rate of postoperative infections in orthognathic surgery.

Secondary objectives are to state and formulate a consensus in prescribing postoperative antibiotics.

Study Design:

The current study is a prospective, double blind, randomized, placebo control, clinical trial.

The impact of post-operative antibiotics in prevention early surgery related infections will be investigated. The potential benefit of the study lies particular in reducing the various side effects of unwise administration of antibiotics, along with the high cost and bacterial resistant resulted from antibiotics overuse.

The study subjects will be allocated by the investigator into two study groups through the use of randomization. The Intervention group will be getting intra-venous1GR Amoxicillin Clavulanate 3 times a day for 5 days post surgery; while the Control group will be getting intra-venous Placebo for 5 days.

As described above, 50 patients will participate in this study, an important prerequisite for this study is a completely healthy patients. Then the patients will be allocated randomly into two subgroups: intervention group and control group, as mentioned before.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Patients
2. >=18 of age
3. If female, is neither pregnant nor lactating
4. Hemoglobin: >10.5 gm/dl, WBC> 4000mm3, platelets>140.00/mm3
5. Negative to allergic reaction to penicillin (Amoxicillin Clavulanate)
6. Negative to allergic reaction to Natural Rubber Latex
7. No immune depressive drugs, e.g. / corticosteroids, cyclosporine, methotrexate, or anti cancer agents, in past one year. Subjects on topical corticosteroids to treat dermatological conditions covering not more than 5% of body surface area are considered eligible
8. Able to provide informed consent
9. Must have normal immune function

Exclusion Criteria:

1. 18> years of age.
2. Any acute or chronic viral, bacterial, immune or other disease in a state usually associated with abnormal cellular immunity (HIV, hepatitis, lung disease).
3. History of allergic reactions.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-02 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
post operative infection in all patients(50 patients) | three months
  the post operative infection will be evaluated using blood tests ( CRP, and WBC)

IPD SHARING:
Plan to Share IPD: Undecided